CLINICAL TRIAL: NCT06060977
Title: A Phase 1b/2a Study to Evaluate the Safety, Pharmacokinetics and Efficacy of IMG-007 in Adult Alopecia Areata Participants With 50% or Greater Scalp Hair Loss
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics and Efficacy of IMG-007 in Adult Alopecia Areata Participants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inmagene LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMG-007-202
Record Dates: First submitted 2023-09-21; First posted 2023-09-29 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Alopecia Areata (AA)
Keywords: IMG-007; Alopecia Areata; Alopecia; Hair Loss; Skin Disease; Immune System Disorder; Dermatologic Agents
MeSH Terms: conditions — Alopecia Areata; Alopecia; Skin Diseases; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMG-007 Dose 1 (300 mg) (Experimental): IMG-007 Dose 1 (300 mg) will be administered intravenously 3 times over 4 weeks
  Interventions: Drug: IMG-007
- IMG-007 Dose 2 (600 mg) (Experimental): IMG-007 Dose 2 (600 mg) will be administered intravenously 3 times over 4 weeks
  Interventions: Drug: IMG-007

INTERVENTIONS:
Drug: IMG-007 — Intravenous Infusion

SUMMARY:
The primary objective of the study is to evaluate the safety of IMG-007 in adults with Alopecia Areata.

DETAILED DESCRIPTION:
This is a phase 1b/2a, open label study to assess the safety, PK, and efficacy of IMG-007 in adult AA participants with 50% or greater scalp hair loss. The study will consist of two cohorts with three periods: a screening period of up to 5 -weeks, a 16-week treatment period and a 20-week follow- up period. Approximately 6 and 24 participants will be sequentially enrolled into cohort 1 and cohort 2, respectively, to receive three intravenous infusions of IMG-007 over 4 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged ≥ 18 and ≤ 65 years
* AA with current episode of hair loss of > 6 months but < 8 years
* AA with ≥ 50% scalp involvement as defined as SALT score ≥ 50

Key Exclusion Criteria:

* Known hepatitis B, hepatitis C, or human immunodeficiency virus infection
* Evidence of active or latent tuberculosis (TB)
* History of untreated or inadequately treated TB infection.
* Active infection requiring treatment with systemic antibiotics, antivirals, antifungals, antiparasitics or antiprotozoals at the Screening visit
* Concurrent hair loss due to other etiologies
* Primary "diffuse" type of AA
* Active inflammatory diseases on the scalp that would interfere with the assessment of AA
* History or presence of hair transplants or micropigmentation of the scalp
* Active systemic diseases that may cause hair loss
* Other conditions or laboratory abnormality that could increase the risk associated with study participation or could interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (11):
  - Northwest Arkansas Clinical Trials Center, PLLC/ Hull Dermatology P.A., Rogers, Arkansas
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - Dawes Fretzin Clinical Resarch Group, LLC, Indianapolis, Indiana
  - Options Research Group, West Lafayette, Indiana
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Great Lakes Research Group Inc., Bay City, Michigan
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - Skin Search of Rochester, Inc., Rochester, New York
  - Stride Clinical Research LLC, Sugar Land, Texas
  - Dermatology Specialists of Spokane, Spokane, Washington
- Canada (6):
  - SimcoMed Health Ltd., Barrie, Ontario
  - Skin Health, Cobourg, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - Research Toronto, Toronto, Ontario
  - Centre de Recherche Saint-Louis, Québec, Quebec
  - Innovaderm Research Inc., Montreal

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- IMG-007 300 mg: IMG-007 300 mg will be administered intravenously 3 times over 4 weeks
  IMG-007: Intravenous Infusion
- IMG-007 600 mg: IMG-007 600 mg will be administered intravenously 3 times over 4 weeks
  IMG-007: Intravenous Infusion
Period: Overall Study
Arm/Group | IMG-007 300 mg | IMG-007 600 mg
Started | 6 | 23
Completed | 5 | 23
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMG-007 300 mg | IMG-007 600 mg | Total
Number analyzed (Participants) | 6 | 23 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 23 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The analysis was based on patients who received IMG-007 300 mg, IMG-007 600 mg and Combined IMG-007.
  years | 42.2 (15.51) | 44.7 (15.05) | 44.2 (14.90)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The analysis was based on patients who received IMG-007 300 mg, IMG-007 600 mg and Combined IMG-007.
  Participants
    Female | 6 | 16 | 22
    Male | 0 | 7 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analysis was based on patients who received IMG-007 300 mg, IMG-007 600 mg and Combined IMG-007.
  Participants
    Hispanic or Latino | 0 | 2 | 2
    Not Hispanic or Latino | 6 | 21 | 27
    Unknown or Not Reported | 0 | 0 | 0
Severity of ALopecia Tool (SALT) Score [Mean (Standard Deviation); unit: units on a scale] — The Severity of Alopecia Tool (SALT) is a quantitative assessment of AA severity by the investigator based on scalp terminal hair loss. To evaluate the efficacy of multiple doses of IMG-007 in AA participants as measured by Severity of Alopecia Tool (SALT) on a scale of 0 for no hair loss, and 100 is complete hair loss (higher scores attributes to worse outcomes). Population: The analysis was based on patients who received IMG-007 300 mg, IMG-007 600 mg and Combined IMG-007.
  units on a scale | 87.23 (15.651) | 78.63 (18.401) | 80.41 (17.954)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Adverse Events in Participants
Description: To evaluate adverse events (AEs) emergent from multiple doses of IMG-007 in adult participants with AA.
Time Frame: Adverse events were collected from baseline through the end of the study, a period of up to 24 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | IMG-007 300 mg | IMG-007 600 mg
Number analyzed (Participants) | 6 | 23
Participants
  Participants with at least 1 TEAE | 3 | 19
  SAE | 0 | 0
  TEAE that was an infusion-related reaction | 1 | 0
  TEAE leading to 4-week dosing period discontinuation | 0 | 0
  TEAE with outcome of death | 0 | 0

2. Secondary Outcome: Evaluation of Severity of Alopecia Tool (SALT)
Description: To evaluate the efficacy of multiple doses of IMG-007 in AA participants as measured by the Severity of Alopecia Tool (SALT). The Severity of Alopecia Tool (SALT) is a quantitative assessment of AA severity by the investigator based on scalp terminal hair loss. To evaluate the efficacy of multiple doses of IMG-007 in AA participants as measured by Severity of Alopecia Tool (SALT) on a scale of 0 for no hair loss, and 100 is complete hair loss (higher scores attributes to worse outcomes).
Time Frame: Mean percent change from baseline in Severity of ALopecia Tool (SALT) at week 24.
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | IMG-007 300 mg | IMG-007 600 mg
Number analyzed (Participants) | 6 | 23
percentage of change | -1.07 (7.593) | -14.32 (3.875)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline through the end of the study, a period of up to 24 weeks.
Arm/Group | IMG-007 300 mg | IMG-007 600 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/23
Other Adverse Events (participants affected / at risk) | 2/6 | 8/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMG-007 300 mg (N=6) | IMG-007 600 mg (N=23)
Headache (Nervous system disorders) | 2 | 2
Hypertension (Vascular disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2
Streptococcal infection (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-08-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT06060977/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT06060977/SAP_001.pdf